CLINICAL TRIAL: NCT02742077
Title: CorPath® 200 RAPID II Study (Robotic-Assisted Peripheral Intervention for Peripheral Arterial Disease)
Brief Title: Robotic-Assisted Peripheral Intervention for Peripheral Arterial Disease II
Acronym: RAPID II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corindus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-01
Record Dates: First submitted 2016-04-12; First posted 2016-04-18 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Robotic-assisted PVI (Other): Robotic-assisted peripheral vascular intervention
  Interventions: Device: Robotic-assisted peripheral vascular intervention

INTERVENTIONS:
Device: Robotic-assisted peripheral vascular intervention — Remote delivery and manipulation of guidewires and rapid exchange catheters during percutaneous vascular interventions.

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the CorPath 200 System in the remote delivery and manipulation of guidewires and rapid exchange catheters for use in percutaneous vascular interventions.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single center, non-randomized feasibility study of the CorPath 200 System to examine its performance during complete interventions (DCB, Stenting) of the femoropopliteal arteries and patient outcomes at 30 days.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

* At least 18 years of age;
* Symptomatic disease: presence of critical limb ischemia (including tissue loss or rest pain), or lifestyle-limiting claudication requiring intervention in the femoropopliteal arteries; and
* The subject has been informed of the nature of the study and agrees to its provisions and has provided written informed consent.

Angiographic Inclusion Criteria Femoropopliteal artery lesion(s) with stenosis (>50%) or occlusion of up to 120 mm in length as determined by imaging (MRA or Angio) prior to index interventional procedure.

Exclusion Criteria:

General Exclusion Criteria

If any of the following criteria are met, the subject cannot be enrolled in this study:

* Failure/inability/unwillingness to provide informed consent;
* Target vessel has been previously treated with bypass; or
* Enrolled in concurrent clinical study.

Angiographic Exclusion Criteria

• Target vessel:

* Shows evidence of previous dissection or perforation, or
* Has adjacent acute thrombus; or
* Has a pre-existing target artery aneurysm or perforation or dissection of the target artery prior to initiation of the interventional procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Brodmann, MD, Principal Investigator — Medizinische Universtität Graz
Locations (1):
- Medizinische Univeristät Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Robotic-assisted PVI
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Robotic-assisted PVI
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Region of Enrollment [Number; unit: participants]
  Austria | 20

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success
Description: Defined as <50% residual stenosis in all CorPath 200 System treated lesions at the completion of the interventional procedure in the absence of device-related serious adverse events (SAE).
Time Frame: 72 hours or hospital discharge, whichever comes first.
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic-assisted PVI
Number analyzed (Participants) | 20
Participants | 20

2. Primary Outcome: Adverse Events
Description: No device-related serious adverse events.
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic-assisted PVI
Number analyzed (Participants) | 20
Participants | 0

3. Secondary Outcome: Operator Radiation Exposure Dose
Description: Physician operator radiation exposure as recorded on personal Enterprise Dose Dashboard (EDD; Landauer) dosimeters
Time Frame: Procedure
Measure: Mean (Standard Deviation); unit: μSv
Arm/Group | Robotic-assisted PVI
Number analyzed (Participants) | 20
μSv | 1.9 (2.9)

4. Secondary Outcome: Patient Radiation Exposure Dose
Description: Patient Radiation Dose-area-product (DAP)
Time Frame: Procedure
Measure: Mean (Standard Deviation); unit: Gy•m^2
Arm/Group | Robotic-assisted PVI
Number analyzed (Participants) | 20
Gy•m^2 | 566.7 (391.5)

ADVERSE EVENTS:
Arm/Group | Robotic-assisted PVI
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic-assisted PVI (N=20)
Access-site Hematoma (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No